CLINICAL TRIAL: NCT06956209
Title: A First-in-Human, Open-Label, Multicenter Study Evaluating the Safety and Efficacy of an Implantable Device for Direct Bladder Wall Stimulation in Participants With Lower Urinary Tract Symptoms of Underactive Bladder
Brief Title: Akyva First In Human
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Iota Biosciences, Inc (Industry)
Collaborators: Astellas Pharma Inc (Industry); H&A LifeSciences Pty Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iota-AS-AUS-001
Record Dates: First submitted 2025-04-14; First posted 2025-05-04 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Underactive Bladder
Keywords: Underactive Bladder
MeSH Terms: conditions — Urinary Bladder, Underactive

STUDY DESIGN:
Intervention Model Description: First in human
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Akyva System (Experimental): Participants in the study arm will receive a device called the "Akyva System." The Akyva System is an implantable device intended to electrically stimulate the bladder muscle that controls bladder emptying or urination
  Interventions: Device: Direct Bladder Wall Stimulation

INTERVENTIONS:
Device: Direct Bladder Wall Stimulation — The Akyva System is an implantable device intended to electrically stimulate the bladder muscle that controls bladder emptying or urination

SUMMARY:
The goal of this study is to check if the study device, the Akyva System, is safe to use and to find out if it has any possible side effects. Researchers will see if the study device can help you urinate without the need for catheterization, which involves passing a catheter (small tube) into the bladder, and if there is improvement in the leftover urine amount in your bladder after urinating or trying to urinate.

ELIGIBILITY:
List of Eligibility Criteria apply to both Non-neurogenic and Neurogenic underactive bladder study participants unless otherwise noted.

Inclusion Criteria:

* Are male or female, as assigned at birth, aged ≥ 22 years of age.
* Presents lower urinary tract (LUT) symptoms that have been ongoing for at least the past 90 days prior to consent.
* Is currently performing clean intermittent catheterization (CIC) for urinary retention at a rate of ≥3 catheterizations per day, as reflected in a 3-day self-catheterization record taken within 180 days prior to consent or a 7-day self-catheterization record collected between day of consent and before the implant procedure.
* Have a post-void residual (PVR) volume ≥ 300 mL as evaluated at least twice within 180 days prior to screening or during screening. NOTE: Individuals unable to void any volume without catheter assistance, i.e. complete retention, are considered to have a PVR equivalent to pre-catheterization volume.
* Have prior history of recurrent urinary tract infection (UTI) with at least two episodes of infection in the past 180 days or currently managing recurrent UTIs with antibiotic medication (e.g. Hiprex).
* Urodynamic measurements consistent with detrusor underactivity. NOTE: Urodynamics performed within the last 365 days prior to consent are acceptable. (1) Bladder contractility index (BCI) < 100 (in Males) (2) Qmax < 15 mL/s and PdetQmax < 20 cmH2O (in Males or Females).
* Are medically fit to withstand abdominal-pelvic surgery under general anesthesia, as evaluated by standard-of-care pre-operative surgical clearance.
* Females of childbearing potential must agree to the use of contraception for the duration of the study
* Are able to understand the risks associated with the study, are willing and able to provide written informed consent prior to any study-related activity, willing and capable of participating in all follow up assessments and willing to undergo all study assessments as described at an approved clinical investigator site.
* Neurogenic Only: Chronic spinal cord injury (>= 6 months post-injury) with sacral/infrascaral (L1 or below) lesions, or mixed lesions associated with neurogenic lower urinary tract dysfunction (NLUTD).

Exclusion Criteria:

* Have or are scheduled for implant of any active implantable medical device (e.g., pacemaker or intrathecal or infusion pump) or have metallic implants/fragments in the abdomen or pelvis (e.g., piercings or hip replacement). Individuals with fully explanted sacral neuromodulation (SNM) or other implantable medical devices may participate. Individuals with implanted and inactive SNM devices may participate.
* Have a documented allergy to tissue contacting Akyva System materials: tecothane, titanium, silicone, epoxy, stainless steel, nickel/cobalt/chromium/molybdenum, polyether ether ketone (PEEK), platinum, iridium, polymethylpentene (TPX), polycarbonate, polyester.
* In the opinion of the Investigator(s), participants who need or are likely to need magnetic resonance imaging (MRI) as part of their routine care for the duration of the study. If MRI is clinically indicated, during or after the study, explant of the Akyva System may be required
* Have hypersensitivity reaction (Types I-IV) to iodine-containing radiographic contrast dyes, or any documented prior severe allergy resulting in anaphylaxis/intubation.
* Have active infection requiring treatment with antibiotics at Screening, unless cleared before Akyva System Surgical Implant (Visit 2).
* Have any history of prior major pelvic or abdominal surgery that would, in the opinion of the Surgical Co-Investigator, increase the risk of injury to abdominal or pelvic organs during the implant procedure.
* Have any history of genitourinary reconstruction surgery or is considering genitourinary reconstruction surgery within the next 24 months.
* Have a significant clinical finding that would, in the opinion of the Surgical Co-Investigator, increase the risk associated with the implant procedure (e.g. ascites, severe inflammatory disease, bleeding or clotting disorder, other interfering devices etc.).
* Have suboptimally controlled Type I or Type II diabetes, as defined by an HbA1C ≥ 7.0%. NOTE: HbA1C results reported within the last 60 days prior to consent are acceptable.
* Have documented renal dysfunction, defined as an estimated glomerular filtration rate (eGFR) ≤ 50 mL/min/1.73 m² or evidence of hydronephrosis on renal ultrasound or CT urogram. NOTE: Renal function panel and renal ultrasound or CT urograms performed within the last 365 days prior to consent are acceptable.
* Have any history of dialysis or kidney transplant.
* Have a history of kidney or bladder stones within the last 5 years.
* Have any history of bladder cancer.
* Have any history of pelvic cancer diagnosis (e.g. uterine, ovarian, rectal), unless disease-free for ≥ 2 years measured from the day of consent.
* Have any history of radiation cystitis.
* Have locally advanced malignancy or metastatic disease within the past five (5) years from the day of consent, with the exception of adequately treated or cured malignancy with no evidence of disease.
* Non-Neurogenic only: Have had botulinum toxin injection in the bladder or pelvic floor in the past 6 months measured from the day of consent.
* Have any history of major bladder reconstructive surgeries.
* Have a bladder compliance < 20 mL/cmH2O measured during urodynamic study. NOTE: Urodynamic performed within the last 365 days prior to consent are acceptable.
* Non-Neurogenic only: Have a current underlying diagnosis of neurogenic bladder.
* Have any history of an overactive bladder or LUT symptoms suggestive of an overactive bladder.
* Non-neurogenic only: Have an iatrogenic cause of UAB symptoms in the opinion of the PI.
* Currently using an indwelling (e.g. Foley) catheter for bladder emptying, with an exception for nighttime-only use.
* Currently using suprapubic catheters, unless the suprapubic catheter is removed at least 30 days prior to implant
* Females who have had any prior abdominal sacrocolpopexy procedure for pelvic organ prolapse.
* Males with history of elevated PSA or prostate cancer undergoing further evaluation or treatment.
* Participants who are unable to discontinue anticoagulant therapy for the implant procedure.
* Females of childbearing potential who are pregnant, not using medical birth control or who are planning to become pregnant during the anticipated study period.
* Predicted life expectancy of less than one year from the day of consent.
* Have any history of diagnosis of bladder outlet obstruction secondary to bladder neck stenosis, BPH or urethral stricture disease. Participants with prior surgical treatment of BPH with no clinical evidence of obstruction and do not require routine MRI may be included
* Any condition that, in the Investigator's opinion, would preclude participation in the study (e.g., have a medical condition that may interfere with interpretation of study results, inability to adhere to the visit schedule, poor cognitive abilities, poor compliance with treatment regimen, or poor dexterity to use the system etc.).
* Previously (within 5.5x the terminal half-life (drug trial) or 8 weeks (device trial) of the screening visit) or currently enrolled in another investigational drug or device trial.
* Vulnerable persons such as prisoners, mentally-disabled or cognitively impaired, homeless or economically disadvantaged, nursing home patients, or others requiring legally authorized representatives.
* Participants that work in an environment with exposures to high levels of electromagnetic interference such as working with high powered electrical equipment.
* Neurogenic Only: Have any history of sphincterotomies
* Neurogenic Only: Have untreated overactive bladder

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
To characterize the safety of implantation and use of the Akyva System | From enrollment to the end of the treatment at 18 months
  Justification of Endpoint: As this is a first-in-human study, the primary objective is to assess the safety of the implantation and use of the Akyva System for bladder wall stimulation.
  o Treatment-emergent incidence rates of AEs, ADEs, SAEs, SADEs, and UADEs that are procedure- or device-related
To characterize the safety of implantation and use of the Akyva System | From enrollment to the end of the treatment at 18 months
  Justification of Endpoint: As this is a first-in-human study, the primary objective is to assess the safety of the implantation and use of the Akyva System for bladder wall stimulation.
  o No ≥ 20% decrease in eGFR from baseline.

SECONDARY OUTCOMES:
To assess the effect of bladder wall stimulation on bladder emptying | From enrollment to the end of the treatment at 18 months
  Justification of Endpoint: This would be assessed by decrease in residual urine/increase in voiding efficiency or decreases in catheter reliance.
  Partial retention participants, Endpoint is considered successful if one or all of the following criteria are met:
  * Decrease in mean number of daily catheterizations ≥ 50% from pre- implant to post-implant as recorded in the bladder diary
  * Decrease in the mean PVR urine volume during catheter-free voiding ≥ 50% from pre-implant to post-implant with stimulation
  * Increase in voiding efficiency by a factor of 1.5 during catheter-free voiding from pre-implant to post-implant with stimulation
  Complete retention participants, Endpoint is considered successful if one or all of the following criteria are met:
  * Decrease in mean number of daily catheterizations ≥ 50% from pre- implant to post-implant as recorded in the bladder diary
  * ≥ 50% bladder volume voided with stimulation
To assess the surgical feasibility of the Akyva system implantation procedure | From enrollment to the end of the treatment at 18 months
  Justification of Endpoint: Although the surgical approach to accessing the anterior bladder wall is common in practice, the placement and use of the Akyva IPG and Leads is unique. This endpoint aims to analyze the feasibility of the Akyva implantation.
  * Two Akyva Leads sutured to the anterior bladder wall connected to the Akyva IPG, and an Akyva systems check demonstrating functionality verified with no non-compliant errors.

CONTACTS AND LOCATIONS:
Overall Officials: Carmela Cusumano, MS, CCRP, CMDA, Study Director — Iota Biosciences; Mike Woods, MD, Study Chair — iota Biosciences
Locations (2):
- Australia (2):
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland

IPD SHARING:
Plan to Share IPD: Undecided